CLINICAL TRIAL: NCT02476409
Title: Tolvaptan Treatment to Reverse Worsening Outpatient Heart Failure: Possible Role of Copeptin In Identifying Responders (TROUPER)
Brief Title: Tolvaptan For Worsening Outpatient Heart Failure: Role of Copeptin In Identifying Responders
Acronym: TROUPER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-0472
Record Dates: First submitted 2015-06-12; First posted 2015-06-19 (Estimated); Results first posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Congestive Heart Failure
Keywords: congestive heart failure; tolvaptan; copeptin
MeSH Terms: conditions — Heart Failure; Diabetes Insipidus | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tolvaptan (Experimental): Augmentation of current dose of loop diuretic + 30 mg of oral tolvaptan daily
  Interventions: Drug: tolvaptan
- Placebo (Placebo Comparator): Augmentation of current dose of loop diuretic
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: tolvaptan — Study will test the addition of tolvaptan to augmentation of loop diuretic as standard of care for outpatients presenting with worsening heart failure.
  Other Names: Samsca
  Arms: Tolvaptan
Other: Placebo — Placebo for tolvaptan
  Arms: Placebo

SUMMARY:
Patients who present to clinic or in the outpatient setting with worsening heart failure represent a unique opportunity for novel approaches to decongestion (removing fluid) that may more rapidly improve fluid status and symptoms as well as reduce the risk of hospitalization.

In these patients with less severe congestion (fluid overload), combining the vasopressin antagonist tolvaptan with loop diuretics (or fluid pills like furosemide/bumetanide/torsemide) may represent a more effective strategy for decongestion. In addition, looking at patients' copeptin levels may help identify those who are more likely to respond to tolvaptan.

DETAILED DESCRIPTION:
This study will be a randomized, double blind, positive control, multi-center clinical trial enrolling patients who present in the outpatient setting with signs and symptoms consistent with worsening congestive heart failure. The sample size for the study is 40 patients. Candidates for the study will be identified by screening outpatients presenting with worsening heart failure.

Patients who qualify for the study will be enrolled within 24 hours of identification. Patients will be randomized in a 1:1 fashion to one of two treatment arms:

* Augmentation of current daily dose of oral loop diuretic + 30 mg of oral Tolvaptan daily
* Augmentation of current daily dose of oral loop diuretic + placebo of oral Tolvaptan daily

Patients will initiate study medication in a hospital setting and will be observed for a period of time that will depend upon their baseline serum sodium and response to study drug. In most cases patients will be observed for 8 hours. Following this observational period, patients will leave the hospital setting and the remainder of the study will consist of follow-up by outpatient visits or by telephone. All patients will have Day 30 follow up phone contact for assessment of vital status, adverse events and morbidity during this period.

The primary objective of this study will be to compare the effects of oral tolvaptan plus augmented loop diuretic versus augmented loop diuretic on short term changes in body weight with and without stratification for baseline copeptin.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Presenting to clinic with worsening heart failure due congestion (fluid overload) Patient reported worsening fluid overload based on perception of edema and/or weight gain With at least one of the following symptoms

  * Worsening dyspnea on exertion or fatigue
  * Worsening orthopnea or paroxysmal nocturnal dyspnea (PND)
  * Perception of abdominal and/or lower extremity edema
  * Early satiety and/or decreased appetite And at least one of the following signs
  * Lower extremity edema
  * Ascites
  * Elevated jugular venous distension (JVD)
  * Pulmonary rales
* Daily oral dose of loop diuretic
* Prior history of heart failure with this diagnosis for at least 1 month with preserved or reduced left ventricular ejection fraction
* Signed informed consent

Exclusion Criteria:

* Patients with symptomatic hyponatremia will be excluded from the study.
* Patients with severe hyponatremia, defined as serum sodium < 125 milliequivalents per Liter (mEq/L) at the time of screening, will be excluded regardless of whether they are symptomatic or not.
* Patients with the following predisposing factors for osmotic demyelinating syndrome (ODS), assessed by the study investigator judgment, will be excluded: chronic alcoholism at the time of study, severe liver disease, marked malnutrition, and risk for chronic hypoxia.
* Patients currently undergoing renal replacement therapy
* Planned hospitalization for acute heart failure
* History of primary significant liver disease or acute hepatic failure, as defined by the investigator
* Hemodynamically significant arrhythmias
* Acute coronary syndrome (ACS) or acute myocardial infarction within 4 weeks prior to study entry
* Active myocarditis
* Hypertrophic obstructive, restrictive, or constrictive cardiomyopathy
* Severe stenotic valvular disease amendable to surgical treatment
* Complex congenital heart disease
* Constrictive pericarditis
* Clinical evidence of digoxin toxicity
* History of adverse reaction or clinical contraindication to tolvaptan

  * Concomitant use of strong cytochrome P450 3A4 (CYP3A4) inhibitors
  * Inability of patient to sense and/or respond to thirst
  * History of hypersensitivity to tolvaptan
  * Patient is anuric
* Enrollment or planned enrollment in another randomized clinical trial during the study period
* Pregnant or breast-feeding
* Inability to comply with planned study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirkwood F Adams, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gheorghiade M, Gattis WA, O'Connor CM, Adams KF Jr, Elkayam U, Barbagelata A, Ghali JK, Benza RL, McGrew FA, Klapholz M, Ouyang J, Orlandi C; Acute and Chronic Therapeutic Impact of a Vasopressin Antagonist in Congestive Heart Failure (ACTIV in CHF) Investigators. Effects of tolvaptan, a vasopressin antagonist, in patients hospitalized with worsening heart failure: a randomized controlled trial. JAMA. 2004 Apr 28;291(16):1963-71. doi: 10.1001/jama.291.16.1963. PMID 15113814
- [Background] Gheorghiade M, Konstam MA, Burnett JC Jr, Grinfeld L, Maggioni AP, Swedberg K, Udelson JE, Zannad F, Cook T, Ouyang J, Zimmer C, Orlandi C; Efficacy of Vasopressin Antagonism in Heart Failure Outcome Study With Tolvaptan (EVEREST) Investigators. Short-term clinical effects of tolvaptan, an oral vasopressin antagonist, in patients hospitalized for heart failure: the EVEREST Clinical Status Trials. JAMA. 2007 Mar 28;297(12):1332-43. doi: 10.1001/jama.297.12.1332. Epub 2007 Mar 25. PMID 17384438
- [Background] Pang PS, Konstam MA, Krasa HB, Swedberg K, Zannad F, Blair JE, Zimmer C, Teerlink JR, Maggioni AP, Burnett JC Jr, Grinfeld L, Ouyang J, Udelson JE, Gheorghiade M; Efficacy of Vasopressin Antagonism in Heart Failure Outcome Study with Tolvaptan (EVEREST) Investigators. Effects of tolvaptan on dyspnoea relief from the EVEREST trials. Eur Heart J. 2009 Sep;30(18):2233-40. doi: 10.1093/eurheartj/ehp253. Epub 2009 Jun 27. PMID 19561338
- [Background] Konstam MA, Gheorghiade M, Burnett JC Jr, Grinfeld L, Maggioni AP, Swedberg K, Udelson JE, Zannad F, Cook T, Ouyang J, Zimmer C, Orlandi C; Efficacy of Vasopressin Antagonism in Heart Failure Outcome Study With Tolvaptan (EVEREST) Investigators. Effects of oral tolvaptan in patients hospitalized for worsening heart failure: the EVEREST Outcome Trial. JAMA. 2007 Mar 28;297(12):1319-31. doi: 10.1001/jama.297.12.1319. Epub 2007 Mar 25. PMID 17384437
- [Background] Morgenthaler NG, Struck J, Jochberger S, Dunser MW. Copeptin: clinical use of a new biomarker. Trends Endocrinol Metab. 2008 Mar;19(2):43-9. doi: 10.1016/j.tem.2007.11.001. PMID 18291667
- [Background] Szinnai G, Morgenthaler NG, Berneis K, Struck J, Muller B, Keller U, Christ-Crain M. Changes in plasma copeptin, the c-terminal portion of arginine vasopressin during water deprivation and excess in healthy subjects. J Clin Endocrinol Metab. 2007 Oct;92(10):3973-8. doi: 10.1210/jc.2007-0232. Epub 2007 Jul 17. PMID 17635944
- [Background] Morgenthaler NG, Struck J, Alonso C, Bergmann A. Assay for the measurement of copeptin, a stable peptide derived from the precursor of vasopressin. Clin Chem. 2006 Jan;52(1):112-9. doi: 10.1373/clinchem.2005.060038. Epub 2005 Nov 3. PMID 16269513

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tolvaptan | Placebo
Started | 19 | 21
Completed | 19 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolvaptan | Placebo | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 15 | 21
  >=65 years | 13 | 6 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8.9) | 60 (14) | 63 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 13 | 10 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 19 | 20 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 12 | 25
  White | 6 | 9 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 21 | 40
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: percent ejection fraction (%)] | 32 (13) | 34 (18) | 33 (16)
Heart Failure Reduced Ejection Fraction (≤ 40) [Count of Participants; unit: Participants] | 13 | 13 | 26
Edema [Count of Participants; unit: Participants] | 17 | 18 | 35
Dyspnea [Count of Participants; unit: Participants] | 18 | 21 | 39
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.7 (0.8) | 1.4 (0.6) | 1.6 (0.7)
Serum Sodium [Mean (Standard Deviation); unit: mEq/L] | 140 (3.7) | 138 (3.8) | 139 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight at 48 Hours
Description: The primary endpoint for the study will be change in body weight between patients randomized to tolvaptan versus placebo from baseline to 48 hours
Time Frame: Baseline, Day 3 (48 hours)
Population: One participant in the Tolvaptan group missed study Visit 2 (Day 3 (48 hours)) due to adverse weather. This participant subsequently attended study Visit 3 (Day 8) to complete the study. Thus data were available on 18 of the 19 patients in the Tolvaptan group for this endpoint at study Visit 2 (Day 3 (48 hours)).
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 18 | 21
pounds | -3.3 (4.4) | -0.8 (3.5)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; Test type: Superiority; p = 0.094, Kruskal-Wallis

2. Primary Outcome: Change in Body Weight at 48 Hours Stratified by Copeptin
Description: The primary endpoint for the study will be change in body weight between patients randomized to tolvaptan versus placebo from baseline to 48 hours with stratification for baseline copeptin level
Time Frame: Baseline, Day 3 (48 hours)
Population: One participant in the High Copeptin - Tolvaptan group missed study Visit 2 (Day 3 (48 hours)) due to adverse weather. Thus data were available on 11 of the 12 patients in the High Copeptin - Tolvaptan group for this endpoint.
Measure: Mean (Standard Deviation); unit: pounds
Groups:
- High Copeptin - Tolvaptan: High Copeptin (≥ 20 pmol/L) Tolvaptan (augmentation of current dose of loop diuretic + 30 mg of oral tolvaptan daily)
  Tolvaptan: Study will test the addition of tolvaptan to augmentation of loop diuretic as standard of care for outpatients presenting with worsening heart failure.
- High Copeptin - Placebo: High Copeptin (≥ 20 pmol/L) Placebo (augmentation of current dose of loop diuretic)
  Placebo: Placebo for tolvaptan
- Low Copeptin - Tolvaptan: Low Copeptin (< 20 pmol/L) Tolvaptan (augmentation of current dose of loop diuretic + 30 mg of oral tolvaptan daily)
- Low Copeptin - Placebo: Low Copeptin (< 20 pmol/L) Placebo (augmentation of current dose of loop diuretic)
  Placebo: Placebo for tolvaptan
Arm/Group | High Copeptin - Tolvaptan | High Copeptin - Placebo | Low Copeptin - Tolvaptan | Low Copeptin - Placebo
Number analyzed (Participants) | 11 | 12 | 7 | 9
pounds | -2.9 (5.3) | 0.3 (3.7) | -3.8 (3.0) | -2.4 (2.7)
Statistical Analysis 1: Comparison: High Copeptin - Tolvaptan vs High Copeptin - Placebo; Test type: Superiority; p = 0.166, Kruskal-Wallis
Statistical Analysis 2: Comparison: Low Copeptin - Tolvaptan vs Low Copeptin - Placebo; Test type: Superiority; p = 0.491, Kruskal-Wallis

3. Secondary Outcome: Changes in Visual Analog Scale - Patient Dyspnea
Description: Changes in patient reported dyspnea scale from baseline to 48 hours based on the visual analog scale.
  Visual Analog Scale (VAS) - Patient Dyspnea has a minimum value of 0 and a maximum value of 100. Higher scores mean a better outcome.
Time Frame: Baseline, Day 3 (48 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 18 | 21
score on a scale | 21 (23) | 15 (22)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; P-value for Change in Dyspnea VAS - Baseline to Day 3 Tolvaptan versus placebo; Test type: Superiority; p = 0.543, Kruskal-Wallis

4. Secondary Outcome: Change in Loop Diuretic Dose (Furosemide Milligram Equivalents) at 48 Hours
Description: Change in loop diuretic dose at 48 hours where doses of loop diuretic are expressed as furosemide milligram equivalents based on standard conversions of bumetanide and torsemide doses to milligram equivalents of furosemide. The formula for the conversion of doses of loop diuretics were standardized to milligram equivalents of furosemide based on 40 milligrams of furosemide for each 1 milligram of bumetanide and 2 milligrams of furosemide for each 1 milligram of torsemide.
Time Frame: Day 3 (48 hours)
Measure: Mean (Standard Deviation); unit: furosemide milligram equivalents
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 19 | 21
furosemide milligram equivalents | -57 (94) | -11 (79)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; Test type: Superiority; p = 0.050, Kruskal-Wallis

5. Secondary Outcome: Number of Participants With a Decrease in Loop Diuretic Dosing at 48 Hours
Description: Number of participants with a decrease in loop diuretic diuretic dosing at 48 hours in the Tolvaptan group and the Placebo group.
Time Frame: Day 3 (48 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 19 | 21
Participants | 9 | 4
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; Test type: Superiority; p = 0.092, Fisher Exact

6. Secondary Outcome: Change in Loop Diuretic Score Defined Based on Change in Loop Diuretic Use
Description: Change in loop diuretic score defined by change in loop diuretic use at Visit 2. The change in loop diuretic score endpoint was calculated as follows: patients having an increase in loop diuretic use at Visit 2 were given a score of 2, patients with no change a score of 0, and patients with a decrease in loop use at Visit 2 were given a score of -1. Increases in loop diuretic use were given a higher weighting to account for their reflection of treatment failure.
Time Frame: Day 3 (48 hours)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 19 | 21
units on a scale | -0.47 (0.51) | 0 (0.77)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; Test type: Superiority; p = 0.034, Kruskal-Wallis

7. Secondary Outcome: Change in Body Weight at Day 8
Description: Change in body weight at 8 days will be analyzed in a similar fashion to the change in body weight at 48 hours
Time Frame: Baseline, 8 days
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 19 | 20
pounds | -1.8 (3.5) | -2.8 (4.4)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; Test type: Superiority; p = 0.643, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the 30 day study period
Description: Systematic assessment was performed by a combination of methods consisting of standard questionnaires, regular investigator assessment, and regular laboratory testing
Arm/Group | Tolvaptan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 6/19 | 4/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolvaptan (N=19) | Placebo (N=21)
Volume Depletion (Cardiac disorders) | 1 (1) | 1 (1) — Loss of fluid leading to symptomatic volume depletion
Worsening Heart Failure (Cardiac disorders) | 4 (4) | 3 (3) — Worsening signs and symptoms of heart failure requiring hospitalization
Chronic Obstructive Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Chronic Obstructive Lung Disease Exacerbation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT02476409/Prot_SAP_000.pdf